CLINICAL TRIAL: NCT00100685
Title: Phase 2 Open-Label Study of Volociximab (M200) in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Study of M200 (Volociximab) in Patients With Metastatic Renal Cell Carcinoma (RCC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M200-1204; NCT00103077 (obsolete NCT alias)
Record Dates: First submitted 2005-01-04; First posted 2005-01-05 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Renal Cell Carcinoma; Metastases
Keywords: Kidney; renal; cancer; carcinoma; cell; metastatic; metastatic renal cell carcinoma; RCC
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis; Neoplasms; Carcinoma | interventions — volociximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Volociximab administered intravenously at a dose of 10 mg/kg qowk
  Interventions: Drug: Volociximab (anti-α5β1 integrin monoclonal antibody)
- Arm 2 (Experimental): Volociximab administered intravenously at a dose of 15 mg/kg qwk
  Interventions: Drug: Volociximab (anti-α5β1 integrin monoclonal antibody)

INTERVENTIONS:
Drug: Volociximab (anti-α5β1 integrin monoclonal antibody) — Volociximab intravenously (Cohort 1: 10 mg/kg every other week or Cohort 2: 15 mg/kg once a week) for up to 104 weeks or until disease progression, whichever occurs first.

SUMMARY:
This clinical trial is being conducted to determine tumor response and preliminary safety of a monoclonal antibody that specifically binds to a cell surface receptor (α5β1 integrin) and is required for the establishment of new blood vessels during tumor growth, a process known as angiogenesis.

ELIGIBILITY:
Inclusion Criteria

* Males and females of at least 18 years of age with metastatic RCC of predominantly clear cell histology who have received 0 to 2 prior treatment regimens for metastatic disease.
* Measurable disease according to Response Criteria for Solid Tumors.
* Negative pregnancy test (women of childbearing potential only).
* Pretreatment laboratory levels that meet specific criteria.
* Signed and dated informed consent and authorization to use protected health information (in accordance with national and local patient privacy regulations
* Patients must have failed at least one approved or investigational tyrosine kinase inhibitor (TKI).

Exclusion Criteria

* Any of the following histologies of RCC: papillary, chromophobe, collecting duct, or unclassified.
* Known sensitivity to murine proteins or chimeric antibodies or other components of the product.
* Use of any investigational drug within 4 weeks prior to screening or 5 half-lives of the prior investigational drug (whichever is longer).
* Systemic chemotherapy, immunotherapy, radiation therapy, or monoclonal antibody therapy within 4 weeks of M200 administration.
* Documented central nervous system (CNS) tumor or CNS metastasis.
* History of thromboembolic events and bleeding disorders within the past year.
* Medical conditions that may be exacerbated by bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with a confirmed tumor response at any time during the study | Any time during the study

SECONDARY OUTCOMES:
Time to disease progression | Up to 104 weeks
Duration of tumor response | Up to 104 weeks
Pharmacokinetics (PK) of M200 | Day 0 through Study Termination
Immunogenicity | Day 0 through Study Termination

CONTACTS AND LOCATIONS:
Overall Officials: Mihail Obrocea, MD, Study Director — Abbott
Locations (3):
- United States (3):
  - Site Reference ID/Investigator# 70400, Los Angeles, California
  - Site Reference ID/Investigator# 70401, New York, New York
  - Site Reference ID/Investigator# 70399, Cleveland, Ohio